CLINICAL TRIAL: NCT03061539
Title: Nivolumab and Ipilimumab Treatment in Prostate Cancer With an Immunogenic Signature
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-935
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Immunogenic signature
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Two-arm non-randomised, non-comparative phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab & Ipilimumab - Cohort 1 (Experimental): Patients will receive Nivolumab 1 mg/kg + ipilimumab 3 mg/kg every three weeks for a maximum of 4 doses followed by a 6 week gap after last combination dose. The patients will then receive 480 mg flat dose of nivolumab every 4 weeks for up to one year, or until progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Nivolumab & Ipilimumab
- Nivolumab & Ipilimumab - Cohort 2 (Experimental): Patients will receive Nivolumab 3 mg/kg + ipilimumab 1 mg/kg every three weeks for a maximum of 4 doses followed by a 3 week gap after last combination dose. The patients will then receive 480 mg flat dose of nivolumab every 4 weeks for up to one year, or until progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Nivolumab & Ipilimumab

INTERVENTIONS:
Drug: Nivolumab & Ipilimumab — Combination Therapy: Cohort 1: Nivolumab 1 mg/kg + ipilimumab 3 mg/kg every 3 weeks for a maximum of 4 cycles . Cohort 2 : Nivolumab 3mg/kg + ipilimumab 1mg/kg every 3 weeks for a maximum of 4 cycles.
  Treatment free gap after last combination dose : Cohort 1: 6 weeks; Cohort 2: 3 weeks
  Monotherapy: 480 mg flat dose of nivolumab every 4 weeks for up to 10 cycles, or until progression, unacceptable toxicity or withdrawal of consent

SUMMARY:
The primary objective is to test the following hypothesis: Patients with metastatic castrate resistant prostate cancer that have progressed following at least one line of therapy and have an immunogenic signature will respond to combined PD-1 and CTLA4 inhibition.

DETAILED DESCRIPTION:
This is a two-arm non-randomised, non-comparative phase II trial designed to assess the efficacy of nivolumab + ipilimumab in patients with metastatic castrate resistant prostate cancer that have progressed following at least 1 line of therapy and have an specified immunogenic signature. The immunogenic signature is defined by the presence of at least one of the following:

* Mismatch repair deficiency by IHC
* Defective DNA repair detected by a targeted sequencing panel
* High inflammatory infiltrate defined on multiplexed IHC criteria.

Treatment consists of :

Cohort 1:

* Nivolumab 1 mg/kg + ipilimumab 3 mg/kg every three weeks for a maximum of 4 doses
* 6 week gap after last combination dose
* 480 mg flat dose of nivolumab every 4 weeks for up to one year, or until progression, unacceptable toxicity or withdrawal of consent.

Cohort 2:

* Nivolumab 3 mg/kg + ipilimumab 1 mg/kg every three weeks for a maximum of 4 doses
* 3 week gap after last combination dose
* 480 mg flat dose of nivolumab every 4 weeks for up to one year, or until progression, unacceptable toxicity or withdrawal of consent.

Patients must have ongoing androgen deprivation to maintain serum testosterone < 1.73 nmol/L.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castrate resistant prostate cancer.
* Histologically confirmed prostate adenocarcinoma.
* Patient has archival prostate cancer tissue available or is willing to undergo a new biopsy.
* Immunogenic biomarker positive disease - see Appendix 1 NB patients will be included in the trial if they meet all other eligibility criteria. Analysis of the ImS will take place after registration. Patients who do not have ImS positive disease will be withdrawn from the trial.
* WHO performance status of 0-1.
* Adequate haematological status.
* Adequate liver and renal function.
* Has had 1 or more lines of systemic treatment for mCRPC.
* Documented prostate cancer progression within 6 months prior to screening
* Ongoing androgen deprivation with serum testosterone <1.73 nmol/L.

Exclusion Criteria:

* Any history of autoimmune disease, with the exception of patients with a history of autoimmune-related hyperthyroidism or hypothyroidism who are in remission or on a stable dose of thyroid-replacement hormone.
* Patients with prior allogeneic stem cell or solid organ transplantation.
* Active invasive malignancy in the previous 2 years excluding non-melanoma skin cancer.
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.

(History of radiation pneumonitis in the radiation field is permitted).

* Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Patients with risk factors for bowel perforation.
* History of grade ≥2 peripheral neuropathy.
* Received therapeutic oral or intravenous (IV) antibiotics within 14 days prior to enrolment (Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or COPD) are eligible).
* Patients must not have had systemic corticosteroid therapy (>10mg daily prednisone equivalent) for 14 days prior to study entry, or concomitant use of other immunosuppressive medications. The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e., for adrenal insufficiency), and mineralocorticoids (e.g., fludrocortisone) is allowed.
* Prior treatment with Sipuleucel-T, immune checkpoint targeting agents or other novel immune-oncology agents.
* Administration of a live, attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, unstable arrhythmias, or unstable angina.
* Patients with uncontrolled Type 1 diabetes mellitus. Patients controlled on a stable insulin regimen are eligible.
* Patients with uncontrolled adrenal insufficiency.
* Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Composite response rate | Up to 5 years following the start of treatment
  Patients will be considered as having had a treatment response if any one of the following criteria are satisfied:
  * Radiological response (RECIST 1.1)
  * PSA response ≥50% confirmed by a second PSA test at least 4 weeks later (PCWG3 2016)
  * Conversion of CTC count from ≥5 cells/7.5ml at baseline to <5 cells/7.5ml confirmed by a second CTC test at least 4 weeks later (PCWG3 2016)

SECONDARY OUTCOMES:
Overall survival | From date of registration until the date of first documented date of death from any cause, assessed up to 5 years.
Radiological progression free survival | From registration to objective disease progression or death from any cause, whichever comes first, assessed up to 5 years
PSA progression free survival | From registration to PSA progression free survival assessed up to 5 years
Change in patient reported outcome measures (NCI's PRO-CTCAE) | From registration until 5 years post treatment
Frequency and severity of adverse events | For 24 months post the start of trial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mark Linch, Principal Investigator — University College London Hospitals
Locations (1):
- University College London Hospital, London, United Kingdom